CLINICAL TRIAL: NCT01907711
Title: Clinical Trial, Randomized, Controlled, Parallel, to Evaluate the Effectiveness of Acupuncture as a Treatment in Patients Diagnosed With Chronic Fatigue Syndrome.
Brief Title: Clinical Trial to Evaluate the Effectiveness of Acupuncture as a Treatment in Patients Diagnosed With CFS.
Acronym: AV/AS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Conchita Jimenez Gutierrez, Nurse. Master´s: acupuncture. Master´s: clinical research applied to health sciences, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AV/AS; COIB. PR - 2725/12 (Registry Identifier: COIB. PR - 2725/12)
Record Dates: First submitted 2013-06-27; First posted 2013-07-25 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Fatigue Syndrome.; Muscular Diseases.; Cognitive Impairment; Sleep Disturbances; Pain.
Keywords: Acupuncture.; Fatigue syndrome chronic.; Sleep disturbances.; Pain.; Cognitive impairment.
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Muscular Diseases; Cognitive Dysfunction; Parasomnias; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Acupuncture. (Sham Comparator): That through the center of the guide tube is inserted blunt rod, producing the sensation of a prick in each of the eight points that are not acupuncture points. No intervention is a completely inert as it involves some type of peripheral stimulus, but the technique is closer to a placebo and offers interesting option from a methodologic al point of view showing and ability to mimic real acupuncture The points are not used acupuncture points but are fictional points. The patient should remáis lying prone during the 20 minutes of the session, so the placebo technique remains hidden. Every five minutes the acupuncturist will repeat the action in the corresponding eigh points.
  Interventions: Device: Acupuncture.
- True acupuncture (Active Comparator): The AV is an energy balance treatment with the aim of restoring health and well-being of the patient. Since each patient may have moré than three diagnoses of Traditional Chinese Medicine, will undertake a Major effort of synthesis of acupuncture points for treatment in a session, use the AV 8 - 12 needles, are held in place for 20 minutes with bidirectional rotation of the sleeve needle for one minute every five minutes (a total of four rotations for session). And in the AS 8 tube rod guides with blunt tip for 20 minutes. The same time be devoted to the patients in each treatment group similar, the time requested for the period of pre and post-treatment will be identical in all cases.
  Interventions: Device: Acupuncture.

INTERVENTIONS:
Device: Acupuncture. — Who tried the insertion and manipulation between 8 - 12 needles with guide applied at different points of the body, individually selected and customized, after the insertion, the acupoint stimulation is done through manipulation of de needle sleeve to achieve at each point the sensation known as "De Qi".
  Other Names: Assurance in manufacturing. EN ISO9001.; Registration No.: 60007186 DD 0001.; Notified under No 0197 to the EC Commission.

SUMMARY:
background: The Chronic Fatigue Syndrome (CFS) presents many disturbances multidimensional affect holistically to people who have the disease and current management of fatigue, pain, anxiety, depression and sleep disturbances present in this clinical entity is unsatisfactory.

Hypothesis:

The hypothesis of this essay is to contrast that acupuncture is more useful than placebo.

The investigators suggest the use of a clinical study protocol (PEC), randomized, placebo-controlled, acupuncture technique, aimed at increasing the patient's sense of well-being, relief of pain and stiffness, acupuncture is effective to reduce fatigue, anxiety, depression and sleep disorders in patients diagnosed with CFS.

DETAILED DESCRIPTION:
Headline Goal.

Evaluate the effectiveness of true acupuncture (AV) compared to placebo-acupuncture or sham acupuncture (AS) in improving symptoms of patients diagnosed with CFS.

Specific objectives:

* To assess whether, in patients diagnosed with Chronic Fatigue Syndrome, AV treatment, compared to AS, is associated with a reduction in fatigue as measured by the scale FIS (Fatigue impact Scale).
* Check the reduction of pain in patients diagnosed with CFS, following treatment with AS versus AV as measured by the McGill.
* To verify the decrease in the use of analgesics in patients diagnosed with CFS, after treatment with the AV versus AS, by counting these drugs.
* Evaluate reducing anxiety in patients diagnosed with CFS, following treatment with AS AV against measured by HAD scale.
* Assess whether, in patients diagnosed with CFS, treatment with AV compared to AS, is associated with a reduction in depressive symptoms, as measured by the HAD scale.
* To assess the improvement in sleep quality in patients diagnosed with CFS, after treatment with AV compared to the AS, as measured by the Pittsburgh scale.
* Check the quality improvement of health-related life (HRQOL) in patients diagnosed with CFS, after treatment with AV compared to the AS, as measured by the SF-36 (Short Form-36).

Methodology.

Design.

Pilot clinical trial randomized, parallel group, placebo-controlled simulated acupuncture, single-center, prospective, patient and assessor blind. 1:1 randomized trial, the principal investigator unknown randomization to the time the patient is randomized.

Primary endpoint. Scores on the fatigue impact scale (FIS) after treatment with two acupuncture techniques.

Study population and total number of patients. After signing the informed consent, we included 60 patients diagnosed with CFS, 30 in the intervention group (IG) of real acupuncture and 30 in the control group (CG) of sham acupuncture, applying an individualized treatment plan customized according energy assessment of each patient.

Duration of treatment. 4 months.

Relevance.

This pilot study can demonstrate the effectiveness of acupuncture as a treatment for the symptoms of CFS. The reduction in fatigue, anxiety, depression, pain and reduction in the intake of analgesics with improved sleep quality, after treatment with real acupuncture technique, i results in increased quality of life for the patient suffering from CFS.

Inclusion criteria.

* Patients must meet each of the following criteria for admission to the study:
* Patients of both sexes.
* Aged between 18 and 70 years.
* Patients diagnosed as having chronic fatigue syndrome according to the diagnostic criteria Fukuda.
* Patients who have previously given their informed consent for participation in the study.

Exclusion criteria.

* Patients who have had prior treatment with acupuncture.
* Pregnant or lactating.
* Women of childbearing potential not using an effective contraceptive method according to medical criteria.
* Terminal clinical condition.
* History of allergy and / or hypersensitivity to the acupuncture needles.
* Patients who are on anticoagulant therapy.
* Use of investigational agents not registered in the 30 days prior to study entry.
* Patients who are participating in another clinical trial of the same or different nature in the last 30 days prior to inclusion.
* Any individual who, in the opinion of the investigator, may not be able to follow instructions or make a good filling of the therapeutic regimen.
* Subjects who do not grant written consent to participate in the study.
* Labor litigation for reasons of participation in the clinical trial of CFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet each of the following criteria for admission to the study:
* Patients of both sexes.
* Aged between 18 and 70 years.
* Patients diagnosed as having chronic fatigue syndrome according to the diagnostic criteria Fukuda.
* Patients who have previously given their informed consent for participation in the study.

Exclusion Criteria:

* -Patients who have had prior treatment with acupuncture.
* Pregnant or lactating.
* Women of childbearing potential not using an effective contraceptive method according to medical criteria.
* Terminal clinical condition.
* History of allergy and / or hypersensitivity to the acupuncture needles.
* Patients who are on anticoagulant therapy.
* Use of investigational agents or not registered in the 30 days prior to study entry.
* Patients who are participating in another clinical trial of the same or different nature in the last 30 days prior to inclusion.
* Any individual who, in the opinion of the investigator, may not be able to follow instructions or make a good filling of the therapeutic regimen.
* Subjects who do not grant written consent to participate in the study.
* Labor litigation for reasons of participation in the clinical trial of CFS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Fatigue, asses the scale fatigue FÍS. • Fatigue: Scores on the fatigue impact scale (FIS) after treatment with two acupuncture techniques | one year
  first visit,13 visit, 6 months and 1 year

SECONDARY OUTCOMES:
• Pain scale (McGill) (MPQ) | one year
  first visit, 13th visit, 6 months and one year
Sleep quality (Pittsburgh) scale (PSQI) | one year
  first visit, 13th visit, 6 months and one year
Quality of life scale (ST-36) | one year
  first visit, 13th visit, 6 months and one year
Anxiety and depression scale HAD. | one year
  first visit, 13th visit, 6 months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Jimenez Gutierrez, Nurse, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- HValldhebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Vas J, Mendez C, Perea-Milla E. Acupuncture vs Streitberger needle in knee osteoarthritis - an RCT. BMJ 2004;329:1216-219. Vas J, Modesto M, Aguilar I, Santos-Rey K, Benitez- Parejo N, Rivas-Ruiz F: Effects of acupuncture on patients with fibromyalgia: study protocol of a multicentre randomized controlled trial. Trials 2011;12:59. Wang T, Zhan Q, Xue X, Yeung A. A systematic review of acunpunture and Moxibustion treatment for chronic fatigue syndrome in China. Am J Chin Med 2008;36:1-24. Wang JJ, Song YJ, Wu ZC, Chu XO, Wang XH, Wang XJ, et al. A meta analysis on randomized controlled trials of acupuncture treatment of chronic fatigue syndrome. Zhen Ci Yan Jiu 2009;34:421-8.
- See also: Valle Hebrón institut de recerca.org. Barcelona. Spain. — http://www.vhir.org